CLINICAL TRIAL: NCT00471627
Title: New Type of a Pancreaticojejunostomy - a Pilot Study
Brief Title: New Type of a Pancreaticojejunostomy
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tampere University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R06088
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2008-06-10 (Estimated); Status verified 2008-06

CONDITIONS: Pancreaticojejunostomy After Pancreatic Head Resection
MeSH Terms: interventions — Pancreaticojejunostomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Pancreaticojejunostomy without stiches through the pancreas — The pancreas is cut with knife, without electric cautery and without stay sutures. Bleeding is controlled with 2-3 exactly placed stiches. The pancreatic stump is sunk inside the jejunum, which is tightened around the pancreas with a purse string. A biodegradable stent is left into the pancreatic duct to prevent its occlusion when tightning the purse string.

SUMMARY:
Previously we have demonstrated in animal experiments,that pancreas is extremely vulnerable to handling, reacting with the development of pancreatitis. In human pancreatic surgery, post-operative pancreatitis mediates many other post-operative complications. A new anastomosis was developed to diminish the injury, as being without any stitches going through the pancreas. The aims were to study up to 30 patients as phase one study, with an interim analysis in this open uncontrolled trial after the first few patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo peancreatic head resection

Exclusion Criteria:

* Those who refuse from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-12; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Pancreatic fistula, other complications | One year from operation

SECONDARY OUTCOMES:
Patency of the pancreaticojejunostomy | One year

CONTACTS AND LOCATIONS:
Overall Officials: Isto H Nordback, M.D., Principal Investigator — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland